CLINICAL TRIAL: NCT04412486
Title: An Open Label Trial of Transfusion of COVID-19 Convalescent Plasma (CCP) to Patients With Moderate to Severe COVID-19
Brief Title: COVID-19 Convalescent Plasma (CCP) Transfusion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Gailen D. Marshall Jr., MD PhD (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor-Investigator, Gailen D. Marshall Jr., MD PhD, Vice Chair for Research, Department of Medicine; Director, Division of Allergy, Asthma and Clinical Immunology, University of Mississippi Medical Center
Organization: University of Mississippi Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0137
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: COVID-19 Convalescent Plasma; Coronavirus; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Recipient of COVID-19 Convalescent Plasma (CCP) Transfusion (Experimental): Transfusion of COVID-19 convalescent plasma to participants with serious or life threatening complications from COVID-19 or are at high risk to develop serious complications.
  Interventions: Biological: COVID Convalescent Plasma

INTERVENTIONS:
Biological: COVID Convalescent Plasma — One unit of COVID Convalescent Plasma transfused on Day 0
  Other Names: CCP, COVID-19 Convalescent Plasma

SUMMARY:
This research study evaluates the safety and effectiveness for the use of convalescent plasma transfusion as a treatment option for novel coronavirus SARS-CoV-2 infection (COVID-19). Donors who have recovered from COVID-19 with high antibody levels to the CoV-2 virus will donate plasma at a Mississippi Blood Services facility. Recipients with COIVD-19 who have severe or life threatening conditions will receive plasma from those persons who have recovered from COVID-19.

DETAILED DESCRIPTION:
The research purpose is to evaluate the safety and clinical effectiveness of transfusing one unit of banked plasma obtained from patients who have recovered from the novel coronavirus SARS-C0V-2 infection with high titers of IgG antibody to this virus transfused into patients with severe or at high risk of progressing to severe coronavirus-induced disease (COVID-19).

The research hypothesis is that COVID-19 convalescent plasma (CCP) transfusion improves outcomes in patients with COVID-19.

The use of CCP to treat serious and life threatening COVID-19 has a sound biological as well as clinical rationale to provide virus-specific immune protection in patients unable to produce and/or maintain antiviral antibodies. This treatment protocol is designed primarily to offer a rescue therapy in patients with severe and life threatening disease and explore use in patients for whom a progression to serious disease is likely. Examining the specific antibody responses to the virus in transfused patients if/when they show signs of recovery and comparing these values with those obtained before the transfusion may provide information to design more extensive trials aimed at identifying the best patient population for future use of CCP.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Clinician judged serious or life threatening COVID-19 (or at significant risk to develop serious COVID) manifested by at least one of the following:

   1. Laboratory confirmed diagnosis of SARS-CoV-2 infection
   2. Hypoxia (PaO2/FiO2 <300, Pulse oximetry <93% at rest
   3. Evidence of pulmonary infiltration
   4. Respiratory failure
   5. Sepsis
   6. Multiple organ dysfunction or failure (assessed by SOFA score)
3. Informed consent provided by the patient or legally authorized representative (LAR)

Exclusion Criteria:

1. Greater than 21 days from confirmed COVID-19 diagnosis
2. Receipt of pooled immunoglobulin transfusion in previous 28 days
3. History of prior reaction to transfused blood products
4. Currently enrolled in other drug trials that preclude investigational treatment with CoV-2 convalescent plasma transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Change in PaO2/FiO2 after CCP transfusion. | 3 Days
  Change in pre-transfusion respiratory status compared to Day 3 respiratory status measured by PaO2/FiO2.
Change in pulse oximetry status after CCP transfusion. | 3 Days
  Change in pre-transfusion respiratory status compared to Day 3 respiratory status measured by pulse oximetry.
Change in aO2 after CCP transfusion. | 3 Days
  Change in pre-transfusion respiratory status compared to Day 3 respiratory status measured by aO2.
Change in respiratory rate after CCP transfusion. | 3 Days
  Change in pre-transfusion respiratory status compared to Day 3 respiratory status measured by respiratory rate.
Change in intubation status after CCP transfusion. | 3 Days
  Change in pre-transfusion respiratory status compared to Day 3 respiratory status measured by intubation status.

SECONDARY OUTCOMES:
Change in Sequential Organ Failure Assessment (SOFA). | Days 1, 3, 7, and 28
  Change in SOFA score pre-transfusion to Days 1, 3, 7, and 28 post-transfusion.
Change in 8-point ordinal clinical deterioration scale. | Days 1, 3, 7, and 28
  Change in 8-point ordinal clinical deterioration scale pre-transfusion to Days 1, 3, 7, and 28 post-transfusion. The 8-point ordinal scale measured by: 8-death, 7-ventilation in addition to ECMO, CRRT and/or vasopressor; 6-intubation and mechanical ventilation; 5-non-invasive mechanical ventilation or high flow oxygen 4- supplemental oxygen by mask or nasal cannula; 3- hospitalization without supplemental oxygen; 2- limitation of activities and 1- no limitation of activities, discharge from hospital.
Length of ICU/hospital stay. | Days 1, 3, 7, and 28
  Total length of stay in ICU/hospital.
Development of plasma transfusion reactions. | Days 1, 3, 7, and 28
  Presence of any signs or symptoms of plasma transfusion reactions at Days 1, 3, 7, and 28 post-transfusion.
Development of immune complex disorders. | Days 1, 3, 7, and 28
  Presence of any signs or symptoms of immune complex disorders (fever spike, urticarial lesion, arthralgias, myalgias, hematuria, non IgE-mediated anaphylaxis) at Days 1, 3, 7, and 28 post-transfusion.
Change in anti CoV-2 IgM and IgG levels. | Days 1, 3, 7, and 28
  Change in anti CoV-2 IgM and IgG levels pre-transfusion compared to levels on Days 1, 3, 7, and 28 post-transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D Marshall, Jr., MD, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Syal K. COVID-19: Herd immunity and convalescent plasma transfer therapy. J Med Virol. 2020 Sep;92(9):1380-1382. doi: 10.1002/jmv.25870. Epub 2020 Jul 11. No abstract available. PMID 32281679
- [Background] Xu Z, Li S, Tian S, Li H, Kong LQ. Full spectrum of COVID-19 severity still being depicted. Lancet. 2020 Mar 21;395(10228):947-948. doi: 10.1016/S0140-6736(20)30308-1. Epub 2020 Feb 14. No abstract available. PMID 32066525
- [Background] Luke TC, Kilbane EM, Jackson JL, Hoffman SL. Meta-analysis: convalescent blood products for Spanish influenza pneumonia: a future H5N1 treatment? Ann Intern Med. 2006 Oct 17;145(8):599-609. doi: 10.7326/0003-4819-145-8-200610170-00139. Epub 2006 Aug 29. PMID 16940336
- [Background] Wong SS, Yuen KY. The management of coronavirus infections with particular reference to SARS. J Antimicrob Chemother. 2008 Sep;62(3):437-41. doi: 10.1093/jac/dkn243. Epub 2008 Jun 18. PMID 18565970
- [Background] Mo Y, Fisher D. A review of treatment modalities for Middle East Respiratory Syndrome. J Antimicrob Chemother. 2016 Dec;71(12):3340-3350. doi: 10.1093/jac/dkw338. Epub 2016 Sep 1. PMID 27585965
- [Background] van Griensven J, Edwards T, de Lamballerie X, Semple MG, Gallian P, Baize S, Horby PW, Raoul H, Magassouba N, Antierens A, Lomas C, Faye O, Sall AA, Fransen K, Buyze J, Ravinetto R, Tiberghien P, Claeys Y, De Crop M, Lynen L, Bah EI, Smith PG, Delamou A, De Weggheleire A, Haba N; Ebola-Tx Consortium. Evaluation of Convalescent Plasma for Ebola Virus Disease in Guinea. N Engl J Med. 2016 Jan 7;374(1):33-42. doi: 10.1056/NEJMoa1511812. PMID 26735992
- [Background] Ye Q, Wang B, Mao J. The pathogenesis and treatment of the ;Cytokine Storm' in COVID-19. J Infect. 2020 Jun;80(6):607-613. doi: 10.1016/j.jinf.2020.03.037. Epub 2020 Apr 10. PMID 32283152
- [Background] Jiang S, Hillyer C, Du L. Neutralizing Antibodies against SARS-CoV-2 and Other Human Coronaviruses. Trends Immunol. 2020 May;41(5):355-359. doi: 10.1016/j.it.2020.03.007. Epub 2020 Apr 2. PMID 32249063
- See also: Clinical Trials at UMMC - CCP Transfusion Study — https://umc.edu/clinicaltrials/default.aspx?trialid=10191